CLINICAL TRIAL: NCT00006280
Title: A Phase II Multicenter Randomized Trial of Tobramycin for Inhalation in Young Children With Cystic Fibrosis
Brief Title: A Study of the Safety and Efficacy of Tobramycin for Inhalation in Young Children With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: Inhaled Tobramycin (completed); 1R01DK057755-01 (NIH); M01RR000037 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin; Inhalation

INTERVENTIONS:
Drug: Tobramycin for Inhalation

SUMMARY:
This study's primary goals are to test the safety and effectiveness of Tobramycin for Inhalation (TOBIr) in cystic fibrosis (CF) patients who are between 6 months and 6 years of age. This drug is an antibiotic that is inhaled into the lungs by the patient. It has already been studied and approved by the FDA for treatment of CF patients 6 years and older. Lung fluid will be examined for bacteria before and after the 28-day treatment. The amount of bacteria before and after treatment will be compared. This will indicate whether the antibiotic was effective in killing bacteria in the lungs. Once treatment begins, patients will be monitored every 2 weeks throughout the study (5 exams in 56 days). Half of the patients will receive TOBIr, half will receive a placebo (a substance that looks like TOBIr but contains no medication).

ELIGIBILITY:
Inclusion Criteria:

* Age at least 6 months and less than 6 years
* Diagnosis of cystic fibrosis with 2 clinical features consistent with CF and confirmed by either sweat chloride >= 60 mEq/L (by quantitative pilocarpine iontophoresis) or by genotype with 2 identifiable mutations consistent with CF.
* One throat or sputum microbiology culture positive for Pseudomonas aeruginosa (Pa) within 2 weeks to 12 months prior to screening.
* Informed consent by parent or legal guardian.

Exclusion Criteria:

* History of adverse reaction to anesthesia or sedation.
* History of aminoglycoside hypersensitivity.
* History of unresolved anemia (hematocrit < 30%) or thrombocytopenia (platelet count < 100,000/mm3).
* History of hemoptysis with 30 days prior to screening.
* History of abnormal renal function (serum creatinine > 1.5 times the upper limit of normal for age).
* History of clinically documented chronic hearing loss.
* Administration of any investigational drug within 30 days prior to screening.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98
Dates: Start 2000-02; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wagener, M.D., Principal Investigator — The Children's Hospital; Richard Moss, M.D., Principal Investigator — Stanford University/Lucille Packard Children's Health Services at Stanford; Robert Wilmott, M.D., Principal Investigator — Children's Hospital & Medical Center; Michael Konstan, M.D., Principal Investigator — Rainbow Babies and Children's Hospital; Pamela Zeitlin, M.D., Ph.D., Principal Investigator — Johns Hopkins University; David Waltz, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; George Retsch-Bogart, M.D., Principal Investigator — University of North Carolina, Chapel Hill; Peter Hiatt, M.D., Principal Investigator — Baylor College of Medicine; Ronald Gibson, M.D., Ph.D., Principal Investigator — Children's Hospital Regional Medical Center
Locations (9):
- United States (9):
  - Stanford University/Lucille Packard Children's Health Services at Stanford, Palo Alto, California
  - The Children's Hospital, Denver, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital, Boston, Massachusetts
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Ramsey BW, Pepe MS, Quan JM, Otto KL, Montgomery AB, Williams-Warren J, Vasiljev-K M, Borowitz D, Bowman CM, Marshall BC, Marshall S, Smith AL. Intermittent administration of inhaled tobramycin in patients with cystic fibrosis. Cystic Fibrosis Inhaled Tobramycin Study Group. N Engl J Med. 1999 Jan 7;340(1):23-30. doi: 10.1056/NEJM199901073400104. PMID 9878641